CLINICAL TRIAL: NCT02496533
Title: The Prevalence of Anxiety in Patients Undergoing Radiologic Exam
Brief Title: Patient Anxiety During Radiological Examination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Midwestern Regional Medical Center (Other)
Responsible Party: Principal Investigator, Jessica Kapustin, RN Survivorship, Midwestern Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MRMC14-14
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Massage (No Intervention): Subjects in this arm will complete rate their anxiety by visual analog scale (VAS). Blood pressure, pulse and respiration will be recorded before and after imaging. The anxiety VAS will be repeated after the imaging procedure. Subjects in this arm will not receive the hand massage prior to the imaging procedure.
- Hand Massage (Experimental): Subjects in this arm will complete rate their anxiety by visual analog scale (VAS). Blood pressure, pulse and respiration will be recorded before massage, after massage but before imaging, and after imaging.The subjects will receive hand massage prior to the imaging procedure. The anxiety VAS will be repeated after the imaging procedure.
  Interventions: Procedure: Hand Massage

INTERVENTIONS:
Procedure: Hand Massage — The hand massage procedure comprises 4 minutes of manipulation of the subject's hands (2 minutes per hand) by a skilled massage therapist or appropriately trained staff.
  Arms: Hand Massage

SUMMARY:
This clinical trial design evaluates whether hand massage reduces anxiety levels in cancer patients as they undergo radiological examination to evaluate tumor response. Anxiety levels will be investigated before massage, after massage, and following the completion of the radiological exam. The Visual Analog Scale (VAS), a validated anxiety assessment tool, will be used to measure anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years
* Scheduled to undergo radiologic imaging evaluation of a tumor

Exclusion Criteria:

* Known hand injury within 30 days prior to study participation
* Known pregnancy
* Mental disability as determined by the treating physician
* Actively receiving radiation therapy
* Actively receiving chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kapustin, RN-C, Principal Investigator — Midwestern Regional Medical Center

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hand Massage | No Massage
Started | 105 | 112
Completed | 102 | 106
Not Completed | 3 | 6
Not completed — Lack of data on outcome | 3 | 0
Not completed — Patient did not complete all measures | 0 | 4
Not completed — Late for radiologic testing | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hand Massage | No Massage | Total
Number analyzed (Participants) | 105 | 112 | 217
Age, Customized [Number; unit: participants]
  Age ≥18 years | 105 | 112 | 217
Gender [Count of Participants; unit: Participants]
  Female | 43 | 46 | 89
  Male | 62 | 66 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 99 | 105 | 204
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 20 | 41
  White | 75 | 86 | 161
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 105 | 112 | 217

OUTCOME MEASURES:

1. Primary Outcome: Change in Anxiety as Measured by Visual Analog Scale
Description: Subjects self-reported their perceived anxiety by marking a visual analog scale (VAS). The VAS covers the range 0 to 10. Higher values indicate greater anxiety (worse outcome). Analysis based on difference reported anxiety score between Baseline and after imaging.
Time Frame: Baseline and After Imaging
Population: All patients completing the study per protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hand Massage | No Massage
Number analyzed (Participants) | 102 | 106
units on a scale
  Baseline | 3.4 (3.5) | 2.1 (2.6)
  After Imaging | 1.6 (2.4) | 1.9 (2.5)
Statistical Analysis 1: Comparison: Hand Massage vs No Massage; H0: No difference in reported anxiety as self-reported change of VAS between Baseline and After Imaging time points between the Massage and No Massage groups After Imaging; Test type: Superiority or Other; p < 0.001, ANOVA — No multiple comparisons were conducted in this analysis. P-value not adjusted for multiple comparisons. No interim analyses performed; Mean Difference (Net) = 1.8

2. Secondary Outcome: Change in Blood Pressure in mmHg
Description: A trained clinician will measure and record the subject's blood pressure using standard practices.
Time Frame: Baseline and After Imaging
Population: All patients completing the study per protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hand Massage | No Massage
Number analyzed (Participants) | 102 | 106
mmHg
  Systolic Blood Pressure Baseline | 132.9 (17.6) | 129.9 (19.9)
  Systolic Blood Pressure After Imaging | 135.1 (16.7) | 136.9 (20.4)
  Diastolic Blood Pressure Baseline | 74.9 (10.3) | 75.1 (10.8)
  Diastoloc Blood Pressure After Imaging | 72.6 (10.2) | 74.7 (11.3)
Statistical Analysis 1: Comparison: Hand Massage vs No Massage; H0: No difference in reported systolic blood pressure measurements between Baseline and After Imaging time points between the Massage and No Massage groups After Imaging; Test type: Superiority or Other; p < 0.02, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Hand Massage vs No Massage; H0: No difference in reported diastolic blood pressure between Baseline and After Imaging time points between the Massage and No Massage groups After Imaging; Test type: Superiority or Other; p < 0.09, ANOVA — No multiple comparisons were conducted in this analysis. P-Value not adjusted for multiple comparisons. No interim analyses were performed

3. Secondary Outcome: Change in Respiration Rate in Breaths Per Minute
Description: A trained clinician will measure and record the subject's respiration rate using standard practices.
Time Frame: Baseline and After Imaging
Population: All patients completing the study per protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Hand Massage | No Massage
Number analyzed (Participants) | 102 | 106
breaths per minute
  Respiration Rate Baseline | 17.2 (2.8) | 17.2 (2.5)
  Respiration Rate After Imaging | 16.6 (2.5) | 17.5 (2.4)
Statistical Analysis 1: Comparison: Hand Massage vs No Massage; H0: No difference in reported respiration rate between Baseline and After Imaging time points between the Massage and No Massage groups After Imaging; Test type: Superiority or Other; p < 0.009, ANOVA — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change in Pulse Rate
Description: A trained clinician will measure and record the subject's radial pulse rate using standard practices.
Time Frame: Baseline and After Imaging
Population: All patients completing the study per protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Hand Massage | No Massage
Number analyzed (Participants) | 102 | 106
beats per minute
  Pulse Rate Baseline | 78.3 (14.6) | 80.6 (14.2)
  Pulse Rate After Imaging | 77.0 (14.0) | 80.1 (15.1)
Statistical Analysis 1: Comparison: Hand Massage vs No Massage; H0: No difference in reported pulse rate between Baseline and After Imaging time points between the Massage and No Massage groups After Imaging; Test type: Superiority or Other; p < 0.45, ANOVA — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Hand Massage | No Massage
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/112
Other Adverse Events (participants affected / at risk) | 0/105 | 0/112

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes